CLINICAL TRIAL: NCT06771323
Title: Safety and Effectiveness of Valbenazine as Adjunct Therapy to Botulinum Toxin Injections in Cervical Dystonia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: HM20029848
Record Dates: First submitted 2025-01-08; First posted 2025-01-13 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Cervical Dystonia
MeSH Terms: conditions — Torticollis | interventions — valbenazine

STUDY DESIGN:
Intervention Model Description: Investigator-Initiated prospective double-blind crossover clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomization assignment (protocol biostatistician) will be provided to the pharmacy, who will remain unblinded and dispense study drug. The study team and subject will be blinded to the order of procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo for their initial injection cycle then switch onto Valbenazine for next injections. (Experimental): Subject will receive the placebo for their initial injection cycle (for 3 months) and then switch onto Valbenazine at the time of their next injections.(next 3 months)
  Interventions: Drug: Valbenazine; Drug: Placebo
- Albenazine for the first injection cycle then switch to Placebo for next injections (Experimental): Subject will receive albenazine for the first injection cycle (duration of 3 months) and then switch onto Placebo at the time of their next injections (remain on it for the next 3 months).
  Interventions: Drug: Valbenazine; Drug: Placebo

INTERVENTIONS:
Drug: Valbenazine — To assess if valbenazine 80mg daily improves motor symptoms in idiopathic CD patients with persistent symptoms despite current treated with botulinum toxin injections.
Drug: Placebo — Placebo

SUMMARY:
The most common form of idiopathic dystonia is adult-onset cervical dystonia (CD), a focal form of dystonia affecting the muscles of the neck. CD is often associated with pain and limited range of motion, and frequently leads to reduced quality of life and disability. Effective long-term treatment options are extremely limited. Recurring botulinum neurotoxin (BoNT) injections can ease the symptoms of CD, but they frequently provide only partial relief and can be associated with intolerable side effects. Deep brain stimulation can be used to treat more severe cases of CD, but this neurosurgical procedure is invasive, on average only about 50% effective and may lead to serious adverse effects. Novel treatment approaches for CD are desperately needed to alleviate symptoms and improve the quality of life for the many who suffer from this chronic and disabling neurological disorder.

DETAILED DESCRIPTION:
The dopaminergic system has been implicated in the pathophysiology of hyperkinetic movement disorders including dystonia. For example, it is well established that acute and chronic dystonia syndromes can be caused by dopamine receptor-blocking drugs. Several animal and human imaging studies also support the presence of abnormal dopaminergic function in idiopathic forms of dystonia. Although historically dopamine receptor-blocking medications have been used to treat dystonia, early clinical trials have been limited and the results mixed. The atypical neuroleptic clozapine was found to be moderately effective in treating segmental and generalized dystonia, but its usefulness was limited by potential adverse effects. Another atypical neuroleptic risperidone has been reported to be effective in a 4-week trial of five patients with various forms of dystonia. Dopamine depleting medications such as the VMAT2 inhibitor tetrabenazine has also been found helpful in some patients with dystonia, particularly those with tardive dystonia, which has overlapping phenomenology with idiopathic dystonia. The more recently developed VMAT2 inhibitor valbenazine has demonstrated clear benefit in tardive dyskinesia, but their therapeutic benefit in idiopathic dystonia has not been evaluated in a placebo-controlled clinical trial. Off label uses and an open-label study of valbenazine suggest it could provide some benefit and be well tolerated in idiopathic CD patient populations.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic CD (neck musculature first and most prominently affected)
* 18-75 years old (participants excluded if their dystonia symptoms began before age 18 as childhood-onset dystonia typically represents a genetic and/or primary generalized form of dystonia)
* Onset of dystonia ≥18 years old, no known hyperkinetic movement disorder-related genetic mutation
* Dystonia severity more than minimal and not very severe as defined by Toronto Western Spasmodic Torticollis Rating Scale-2 Motor Severity (TWSTRS-2-Severity) score ≥ 5 and ≤ 20.
* Stable on botulinum toxin injections last 90 days (BoNT dose change <10% and patient reported stability of response over last two injection cycles)
* Stable on other neuroactive medications.

Exclusion Criteria:

* History of deep brain stimulation
* History of uncontrolled or untreated depression in the prior 3 months, suicidality, or history of suicide attempts
* History of uncontrolled liver disease or failure
* History of tardive dyskinesia or tardive dystonia
* Currently taking dopaminergic and/or anti-dopaminergic medications including VMAT2 inhibitors or other antipsychotic medications
* Exposure to dopaminergic and/or anti-dopaminergic medications including VMAT2 inhibitors or other antipsychotic medications in the last 30 days -Presence of parkinsonism or other movement disorder other than dystonia on exam -Receiving botulinum toxin injections at a planned frequency other than every 3 months or typically receive injections at intervals <11 weeks or >13 weeks -Known history of long QT syndrome or cardiac tachyarrhythmia or any clinically significant cardiac abnormality.
* Prolonged QTc as defined by > 450 msec for men and > 470 msec for women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Toronto Western Spasmodic Torticollis Rating Scale-2 (TWSTRS)-severity score change at 12 weeks of treatment | baseline and 12 weeks of treatment
  TWSTRS-2-severity score change at 12 weeks of treatment. The isolated TWSTRS-2-Severity score change was chosen as the primary outcome because the TWSTRS-2-Severity had items dropped from the original TWSTRS as they failed to meet criteria for utility in clinimetric testing,11 and because the primary effect of Valbenazine is expected to be on the motor symptoms and less on pain and disability. The Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS-2) uses the following scoring system for severity:
  0: Absent, 1: Mild, which is less than one-third of the possible range and can be intermittent or constant 2: Moderate, which is one-third to two-thirds of the possible range and constant, or severe, which is more than two-thirds of the possible range and intermittent, and 3: Severe and constant

SECONDARY OUTCOMES:
Global Dystonia Severity Rating Scale (GDSRS) | Visit 2 (Baseline, Week 1) and Visit 3 (Week 6)
  Pain in Dystonia Scale (PIDS), The GDS is a Likert type scale with ratings from 0 to 10 (0 is no dystonia, 1 minimal, 5 moderate and 10 severe dystonia). There are no modifying ratings or weighting factors in the GDS. The total score is the sum of the scores for all the body areas. The maximal total score of the GDS is 140.
Hospital Anxiety and Depression Scale (HADS) | Visit 2 (Baseline, Week 1) and Visit 3 (Week 6)
  It comprises 14 items (7 items each for anxiety and depression), with a score ranging between 0 and 21 for the anxiety and depression subscales. For each subscale the total score is at most 21. A score of ≥11 is considered a clinically significant disorder, whereas a score between 8 and 10 suggests a mild disorder.
Pittsburgh Sleep Quality Index (PSQI) | Visit 2 (Baseline, Week 1) and Visit 3 (Week 6)
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. Scores for each question range from 0 to 3, with higher scores indicating more acute sleep disturbances. Developers have suggested a cut- off score of 5 for the global scale as it correctly identified 88.5% of the patient group in their validation study.
Epworth Sleepiness Scale (ESS) | Visit 2 (Baseline, Week 1) and Visit 3 (Week 6)
  The ESS is a short, self-administered questionnaire designed to measure sleep propensity in a simple, standardized way (only 8 questions on a total scale of 0 to 24).
Cervical Dystonia Impact Profile - 58 item (CDIP-58) | Visit 2 (Baseline, Week 1) and Visit 3 (Week 6)
  A Cervical Dystonia Impact Profile-58 (CDIP-58) score represents a patient's self-reported assessment of how much their cervical dystonia impacts their quality of life, with a higher score indicating a greater negative impact across various aspects like pain, movement limitations, sleep disturbances, mood, and social functioning; essentially, a higher score means a more significant impact from their cervical dystonia. The score is calculated from 58 questions, each rated on a scale, resulting in a total score between 0 (no impact) and 100 (severe impact).
Clinical Global Impression of Severity scale (CGI-S) | Visit 2 (Baseline, Week 1) and Visit 3 (Week 6)
  The Clinical Global Impression Scale-Severity (CGI-S) is a 7-point categorical scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis.The CGI-Severity (CGI-S) asks the clinician one question: "Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?" which is rated on the following seven-point scale: 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4: Moderately ill 5: Markedly ill 6: Severely ill 7: Among the most extremely ill patients
Patient Global Impression of Severity scale (PGI-S) | Visit 2 (Baseline, Week 1) and Visit 3 (Week 6)
  The Patient Global Impression of Severity (PGI-S) scale is a single-item, 6-point, self-administered tool and is used to assess health severity in both health economics evaluation and as an outcome measure in clinical trials in a range of diseases.The highest achievable stage in PGI is Level I, which is for scores 951-1000. In between, an equal width of 50 points has been kept for each Level. In the PGI, Level II means PGI score 901-950, Level III: 851-900, Level IV: 801-850, and so on up to Level IX: 551-600.
Columbia Suicide Severity Rating Scale (C-SSRS) | Visit 2 (Baseline, Week 1) and Visit 3 (Week 6)
  The Columbia-Suicide Severity Rating Scale (C-SSRS) is an assessment tool that. evaluates suicidal ideation and behavior. The scale includes 4 dimensions: hopelessness, suicidal ideation, negative self-evaluation, and hostility. Each of the sub dimensions receives a total score and the sum of all scores gives the overall suicide probability score. Total scores that can be obtained from the scale range from 36 to 144
Pain in Dystonia Scale (PIDS) | Visit 2 (Baseline, Week 1) and Visit 3 (Week 6)
  PIDS offers practicality featuring self-rating of pain intensity using a visual analogue scale, evaluation of pain across body regions, assessment of pain's impact on daily activities, and consideration of external factors that trigger or alleviate pain.The Scale is a 5-point, criterion-based, ordinal scale designed to assess dystonia in eight body regions: eyes, mouth, neck, trunk, and the four extremities (see Appendix I). Raters score dystonia as none (0), slight (1), mild (2), moderate (3), or severe (4).

CONTACTS AND LOCATIONS:
Overall Officials: Brian Berman, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No